CLINICAL TRIAL: NCT05227430
Title: Standardized Educational Videos of Laparoscopic Gynecological Surgeries for the Improvement of Surgical Performance of Surgical Trainees
Brief Title: Standardized Educational Videos of Laparoscopic Gynecological Surgeries
Acronym: AA-GYNLAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Aya Mohr Sasson, Principle investigator, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AA-GYNLAP
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Educational Problems; Surgery; LAP; GYN Disorders
Keywords: educational video; gynecological laparoscopies; hysterectomy; salpingectomy; oophorectomy
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical trainees (Experimental): Surgical trainees that would be given educational video tutorials before entering gynecological laparoscopic surgeries
  Interventions: Other: Educational video tutorials
- Control (No Intervention): Surgical trainees that would not be given educational video tutorials before entering gynecological laparoscopic surgeries

INTERVENTIONS:
Other: Educational video tutorials — Educational video tutorials (Hysterectomy, Bilateral salpingo-oophorectomy, Bilateral salpingectomy)
  Arms: Surgical trainees

SUMMARY:
Owing to coronavirus disease-related social distancing requirements, online education has gained prominence. Surgical trainers consider online videos as a useful teaching aid that maximizes trainees' learning and skill development given the backdrop of time constraints and productivity demands, however, online videos usually do not undergo a peer-review process. Based on these premises the LAP-VEGaS guidelines (LAParoscopic surgery Video Educational GuidelineS), a recommended checklist for production of educational surgical videos, were developed. This study aime to evaluate the impact of educational videos of laparoscopic gynecological surgeries, that were standardized with the LAP-VEGaS, for the improvement of surgical confidence and performance of surgical trainees.

DETAILED DESCRIPTION:
Introduction Owing to coronavirus disease-related social distancing requirements, online education has gained prominence. Surgical trainers consider online videos as a useful teaching aid that maximizes trainees' learning and skill development given the backdrop of time constraints and productivity demands. YouTube has become the most commonly used online resource for educational material among residents, however, online videos usually do not undergo a peer-review process. Moreover, recent studies questioned the educational quality of YouTube laparoscopic hysterectomy videos.

Based on these premises the LAP-VEGaS guidelines (LAParoscopic surgery Video Educational GuidelineS), a recommended checklist for production of educational surgical videos, were developed by an international, multispecialty, joint trainers-trainees committee aiming to reduce the gap between surgeons' expectations and online resources' quality. The LAP-VEGaS VAT is considered valid and practical tool for assessing online laparoscopic operation videos. It assesses nine items. Every item scoring from 0 (item not presented in the video) to 2 (item extensively presented in the video) with a total marking score ranging from 0 to 18. Studies have reported highly accurate in identifying and selecting videos for acceptance for conference presentation and publication, with high level of internal consistency and generalizability. However, the question of how effectively standardized videos serve as quality influencing educational material remains unanswered. Additionally, date regarding its implication in gynecological laparoscopic interventions is limited.

Due to the aforementioned the aim of this study is to evaluate the impact of educational videos of laparoscopic gynecological surgeries, that standardized with the LAP-VEGaS, for the improvement of surgical confidence and performance of surgical trainees.

Material and Methods:

This a prospective study including residents at the beginning of gynecology round in two medical centers. Educational video tutorials of gynecological laparoscopic surgeries (Hysterectomy, Bilateral salpingo-oophorectomy (BSO), Bilateral salpingectomy) will be prepared following the LAP-VEGaS VAT standardization.

Residents in only one medical center will be asked to view the study educational videos (Study group). Residents in the other medical center will not receive the prepared video tutorials and will be free to use other modalities (Controls). Both groups will complete pre-operative questionnaire regarding their subjective self-evaluation of confidence in the stages of the procedures, instrumentation used, anatomy, potential risks and methods to control them. Additional post-operative questionnaire regarding performance during operation, familiarity with operative stages, anatomy and participants will be completed by the senior surgeon evaluating the resident and by all residents participating in the study. Data regarding residents' characteristics will be collected. Groups will be compared for differences in subjective confidence before surgery, performance during surgery and satisfaction rate.

ELIGIBILITY:
Inclusion criteria:

- Residents and fellows in OBGYN in their gynecological round

Exclusion criteria:

- Residents and fellows that did not complete module training for laparoscopic surgeries

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Performance evaluation by senior surgeon | At the end of the operation
  Evaluated by the senior surgeon using the global rating scale of operative performance:7 questions rated between 1 (low performance) to 5(highly skilled)

SECONDARY OUTCOMES:
Performance evaluation- evaluated by the trainee | At the end of the operation
  valuated by the surgical trainee using the global rating scale of operative performance:7 questions rated between 1 (low performance) to 5(highly skilled)

CONTACTS AND LOCATIONS:
Overall Officials: Aya Mohr-Sasson, M.D, Principal Investigator — Aya Mohr-Sasson, Primary Investigator

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Unal F, Atakul N, Turan H, Yaman Ruhi I. Evaluation of YouTube laparoscopic hysterectomy videos as educational materials during the COVID-19 era using the LAParoscopic surgery Video Educational GuidelineS (LAP-VEGaS) and LAP-VEGaS video assessment tool. J Obstet Gynaecol. 2022 Jul;42(5):1325-1330. doi: 10.1080/01443615.2021.1962823. Epub 2021 Oct 27. PMID 34704513
- [Result] Celentano V, Smart N, Cahill RA, Spinelli A, Giglio MC, McGrath J, Obermair A, Pellino G, Hasegawa H, Lal P, Lorenzon L, De Angelis N, Boni L, Gupta S, Griffith JP, Acheson AG, Cecil TD, Coleman MG. Development and validation of a recommended checklist for assessment of surgical videos quality: the LAParoscopic surgery Video Educational GuidelineS (LAP-VEGaS) video assessment tool. Surg Endosc. 2021 Mar;35(3):1362-1369. doi: 10.1007/s00464-020-07517-4. Epub 2020 Apr 6. PMID 32253556
- [Result] Abdelsattar JM, Pandian TK, Finnesgard EJ, El Khatib MM, Rowse PG, Buckarma EN, Gas BL, Heller SF, Farley DR. Do You See What I See? How We Use Video as an Adjunct to General Surgery Resident Education. J Surg Educ. 2015 Nov-Dec;72(6):e145-50. doi: 10.1016/j.jsurg.2015.07.012. Epub 2015 Oct 9. PMID 26454723
- [Result] Celentano V, Smart N, Cahill RA, McGrath JS, Gupta S, Griffith JP, Acheson AG, Cecil TD, Coleman MG. Use of laparoscopic videos amongst surgical trainees in the United Kingdom. Surgeon. 2019 Dec;17(6):334-339. doi: 10.1016/j.surge.2018.10.004. Epub 2018 Nov 9. PMID 30420320
- [Result] Igwe E, Hernandez E, Rose S, Uppal S. Resident participation in laparoscopic hysterectomy: impact of trainee involvement on operative times and surgical outcomes. Am J Obstet Gynecol. 2014 Nov;211(5):484.e1-7. doi: 10.1016/j.ajog.2014.06.024. Epub 2014 Jun 17. PMID 24949539